CLINICAL TRIAL: NCT00663598
Title: REALISE Levitra® - Real Life Safety and Efficacy of Levitra
Brief Title: Levitra® - Real Life Safety and Efficacy of Levitra
Acronym: REALISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100477
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Treatment according to US PI

SUMMARY:
Collect data on safety, efficacy, and subject acceptance of vardenafil treatment under daily life conditions in a large number of subjects with erectile dysfunction (ED)

ELIGIBILITY:
Inclusion Criteria:

* Male outpatients >/= 18 years of age with a diagnosis of ED according to the 1992 US National Institutes of Health (NIH) Consensus Statement (the inability to achieve and maintain penile erection sufficient to complete satisfactory intercourse), and independent of any previous ED treatment

Exclusion Criteria:

* Exclusion according to US PI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30825 (Actual)
Dates: Start 2003-10; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Improvement of Erectile Disfunction | 8 weeks
Onset of Drug Effect | 8 weeks
Second successful intercourse | 8 weeks

SECONDARY OUTCOMES:
General Safety Parameters | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer